CLINICAL TRIAL: NCT03693209
Title: Evaluation of a Brief Intervention Based on Implementation Intentions to Reduce Anger and Aggression in Adolescence: A Randomised Controlled Trial
Brief Title: Using Implementation Intentions to Reduce Anger and Aggression in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Laura Castillo Eito, Principal Investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 017275
Record Dates: First submitted 2018-09-24; First posted 2018-10-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Aggression; Anger
Keywords: Implementation intentions; Volitional Help Sheet; Adolescent
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: There will be one control group and two intervention groups. Each group will be independently be compared with the others, and not in combination.
Who Masked: Participant, Outcomes Assessor
Masking Description: The control condition is active and has a similar format to the intervention conditions to avoid participants knowing which condition they have been assigned to. Outcomes are assessed by self-report.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General trigger (Experimental): VHS with one general trigger: "If I am getting angry..." and 10 strategies (e.g. "Then I will take deep breaths"). Participants are instructed to link trigger with strategies.
  Interventions: Behavioral: Volitional Help Sheet (VHS)
- Specific triggers (Experimental): VHS with a list of 10 specific situations that can act as anger triggers (e.g. "If I am getting angry when people act like they know it all") and 10 strategies. Participants are instructed to link triggers with strategies.
  Interventions: Behavioral: Volitional Help Sheet (VHS)
- Control (No Intervention): List of 10 specific situations that can act as anger triggers and 10 strategies. Participants are instructed to select most encountered triggers and most useful strategies.

INTERVENTIONS:
Behavioral: Volitional Help Sheet (VHS) — VHS with a general anger trigger and 10 anger management strategies
  Other Names: implementation intentions, action-planning
  Arms: General trigger
Behavioral: Volitional Help Sheet (VHS) — VHS with 10 specific anger triggers and 10 anger management strategies
  Other Names: implementation intentions, action-planning
  Arms: Specific triggers

SUMMARY:
This study will test whether making plans of action for situations that trigger anger is effective in reducing anger and aggression in adolescents with behavioural problems.

Participants will be assigned to three groups: a control group and two experimental groups. Participants assigned to the experimental groups will receive either one general anger trigger or a list of specific anger triggers in addition to a list of strategies that can be used to manage anger. Participants will be instructed to link the triggers with the strategies, thus creating action plans with an if-then structure. Participants assigned to the control group will receive the same lists. However, they will receive different instructions which will ask them to select separately the most encountered triggers and the most useful strategies.

It is expected that making plans will reduce the anger and aggression of participants. It is also expected that the reduction will be larger for participants with low violent intentions, low callous-unemotional traits and low impulsivity.

DETAILED DESCRIPTION:
This study aims to test whether aggression in adolescents can be reduced using implementation intentions. This technique involves identifying critical situations that might trigger the unwanted behaviour and making a plan to engage in an alternative course of action when those triggers are present. Implementation intentions formation has been found to be effective in reducing smoking uptake and consultations for emergency contraception in this age group.

A randomised controlled trial will be conducted. Students from 11 to 17 years old attending special schools for children with behavioural problems or referred for anger issues will be randomised to three conditions: attention control, specific triggers and general trigger. Participants in the attention control and specific triggers conditions will receive the same Volitional Help Sheet (VHS), composed of a list of 10 anger triggers (if statements) and a list of 10 anger management strategies (then statements). However, the instructions will be different. Participants in the attention control condition will be instructed to select the triggers that they encounter more often and the strategies that they consider more useful. In contrast, participants in the specific triggers condition will have to link each specific trigger that they encounter often with a specific strategy, thus creating action plans with an if-then structure. Participants assigned to the general trigger condition will also be instructed to make plans linking the trigger with a strategy, but the VHS they will receive will contain only one general trigger: "If I am getting angry".

Measures of anger and reactive physical aggression, reactive relational aggression, proactive physical aggression and proactive relation aggression will be collected at baseline, one month and six months after intervention. In addition, measures of negative urgency, violent intentions and callous-unemotional traits will be collected once.

Both intervention groups are hypothesised to reduce anger and reactive aggression in comparison to the control group. It is hypothesised that the reduction in anger acts as a mediator for the reduction of reactive aggression. It is also hypothesised that violent intentions, callous-unemotional traits and negative urgency act as moderators of effectiveness.

The effects of the intervention will be analysed on anger, on the aggression total score and on the four types of aggression separately using Multivariate Analysis of Covariance. In order to test whether the effect of the interventions on reactive aggression at follow-up is mediated by anger, a mediation analysis will be conducted using the PROCESS macro (Hayes, 2013). In the analysis, the intervention conditions (dummy coded) will be entered as the independent variable, anger as the mediator variable, reactive aggression at follow-up as the dependent variable, and reactive aggression at baseline as the covariate. The analysis will asses the strength of the direct and indirect effects of the interventions on reactive aggression via anger. In order to test whether the effect of the interventions on aggression at follow-up is moderated by violent intentions, callous-unemotional traits and negative urgency, a moderated regression analysis will be conducted using the PROCESS macro (Hayes, 2013). In the analysis, the intervention conditions (dummy coded) will be entered as the independent variable, violent intentions, callous-unemotional traits and negative urgency as the moderator variables, aggression at follow-up as the dependent variable, and aggression at baseline as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Attending a school for children with Social, Emotional and Mental Health needs.
* Being referred by school staff due to anger issues or behavioural problems.

Exclusion Criteria:

* Having severe or profound learning disabilities.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Brief Peer Conflict Scale - Youth self-report (Scott, Lapré, Marsee, & Weems, 2014) | Change from baseline to 6 months after intervention
  Self-report measure of aggression with 20 items. Each item can be rated from 0 (not at all true) to 3 (definitely true). Total scores range from 0 to 60. Higher scores indicate higher aggression. It contains four sub-scales: reactive physical aggression, reactive relational aggression, proactive physical aggression and proactive relational aggression. Each subscale contains 5 items and the score for each range from 0 to 15.

SECONDARY OUTCOMES:
Dimensions of Anger Reactions Scale (DAR-5; Novaco, 1975) | Measured at baseline, one month after intervention and 6 months after intervention
  Self-report measure of anger with 5 items. Each item can be rated from 1 (none or almost none of the time) to 5 (all or almost all of the time). Total scores range from 5 to 25. Higher scores indicate higher anger symptoms.
Peer Conflict Scale - Teacher report (Marsee, Kimonis, & Frick, 2004) | Measured at baseline, one month after intervention and 6 months after intervention
  Teacher report measure of aggression with 40 items. Each item can be rated from 0 (not at all true) to 3 (definitely true). Total scores range from 0 to 120. Higher scores indicate higher aggression. It contains four sub-scales: reactive physical aggression, reactive relational aggression, proactive physical aggression and proactive relational aggression. Each subscale contains 10 items and the score for each range from 0 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Castillo-Eito, Msc, Principal Investigator — University of Sheffield; Christopher J Armitage, PhD, Study Director — University of Manchester; Paul Norman, PhD, Study Director — University of Sheffield; Richard Rowe, PhD, Study Director — University of Sheffield
Locations (3):
- United Kingdom (3):
  - Schools for children with Social Emotional and Mental Health needs., Leeds
  - Schools for children with Social Emotional and Mental Health needs., Sheffield
  - Secondary schools, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scott BG, Lapre GE, Marsee MA, Weems CF. Aggressive behavior and its associations with posttraumatic stress and academic achievement following a natural disaster. J Clin Child Adolesc Psychol. 2014;43(1):43-50. doi: 10.1080/15374416.2013.807733. Epub 2013 Jun 24. PMID 23795776
- [Background] Marsee MA., Kimonis ER., Frick PJ. Peer conflict scale. Unpublished rating scale, University of New Orleans, 2004.
- [Background] Novaco RW. Dimensions of Anger Reactions. Irvine, CA: University of California; 1975.